CLINICAL TRIAL: NCT06062602
Title: TAK-676 Alone and in Combination(s) With Carboplatin, 5-Fluorouracil, and Paclitaxel in Patients With Head and Neck Squamous Cell Carcinoma
Brief Title: PBI-MST-01(NCT04541108) Substudy TAK-02: Intratumoral Microdosing of TAK-676 in HNSCC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Presage Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MST01-TAK-02; PBI-MST-01 (Other: Presage Biosciences)
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC; intratumoral microdosing; microdose injection; microdosing; in vivo oncology; in vivo drug sensitivity; tumor microenvironment; multiplexed immunohistochemistry; head and neck cancer; pharmacodynamic biomarkers; CIVO; master protocol; precision oncology; spatial biology
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Carboplatin; Fluorouracil; Paclitaxel; CP protocol

STUDY DESIGN:
Intervention Model Description: This is an exploratory clinical trial to evaluate intratumoral mechanistic effects of novel and approved agents on intact human tumors. This substudy is not blinded. This is a cohort substudy of a Master Protocol (PBI-MST-01, NCT 04541108) framework that describes the experimental workflow for use of the CIVO platform. Comparisons will not be made between substudy cohorts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAK-676, Carboplatin, 5-FU, & Paclitaxel (Experimental): Patients who are scheduled for surgical biopsy or tumor resection surgery will be injected at least four hours to up to four days prior to surgery using the CIVO device. Each needle of the CIVO device will deliver up to 8.3 microliters of solution, including a vehicle control (sterile saline) or subtherapeutic microdoses of TAK-676, carboplatin, 5-fluorouracil (5- FU), or paclitaxel as single agents or in combination. Each microdose is simultaneously injected in a columnar fashion through each of 8, 5, or 3 needles (in a device configuration determined by tumor dimensions) into a single solid tumor or effaced metastatic lymph node.
  Interventions: Drug: TAK-676; Drug: Carboplatin; Drug: 5-FU; Drug: Paclitaxel; Combination Product: TAK-676 + Carboplatin; Combination Product: Carboplatin + Paclitaxel; Combination Product: Carboplatin + 5-FU; Combination Product: TAK-676 + Carboplatin + 5-FU; Combination Product: TAK-676 + Carboplatin + Paclitaxel

INTERVENTIONS:
Drug: TAK-676 — Intratumoral microdose injection by the CIVO device.
Drug: Carboplatin — Intratumoral microdose injection by the CIVO device.
  Other Names: Paraplatin
Drug: 5-FU — Intratumoral microdose injection by the CIVO device.
  Other Names: Adrucil
Drug: Paclitaxel — Intratumoral microdose injection by the CIVO device.
  Other Names: Taxol
Combination Product: TAK-676 + Carboplatin — Intratumoral microdose injection by the CIVO device.
Combination Product: Carboplatin + Paclitaxel — Intratumoral microdose injection by the CIVO device.
Combination Product: Carboplatin + 5-FU — Intratumoral microdose injection by the CIVO device.
Combination Product: TAK-676 + Carboplatin + 5-FU — Intratumoral microdose injection by the CIVO device.
Combination Product: TAK-676 + Carboplatin + Paclitaxel — Intratumoral microdose injection by the CIVO device.

SUMMARY:
This is a multi-center, open-label Phase 0 substudy designed to study the localized pharmacodynamics (PD) of TAK-676 alone or in combination with Carboplatin, 5-FU, or Paclitaxel within the tumor microenvironment (TME) when administered intratumorally in microdose quantities via the CIVO device in patients diagnosed with Head and Neck Squamous Cell Carcinoma presenting with a surface accessible solid tumor for which there is a scheduled surgical intervention. This substudy is a cohort of the PBI-MST-01 Master Protocol.

DETAILED DESCRIPTION:
CIVO is a research tool composed of a hand-held single-use sterile injector coupled with fluorescent tracking microspheres called CIVO GLO that mark the sites of drug microdose injection, enabling rapid assessment of multiple oncology drugs or drug combinations simultaneously within a patient's tumor. Tumor responses to cancer treatments are highly context-specific and often involve complex interactions between the anti-cancer therapy, genetically diverse tumor cells, and a heterogeneous TME. This complexity is rarely modeled accurately in preclinical translational models of cancer.

In this Phase 0 intratumoral microdosing substudy in human patients with Head and Neck Squamous Cell Carcinoma (who will be undergoing previously planned tumor and/or regional node dissection), we will evaluate the ability of TAK-676 to activate innate immune effector cells within the local tumor microenvironment. Additionally, this study will examine the effect of TAK-676 in combination with Carboplatin, or Paclitaxel, or in combination with 2 agents Carboplatin and 5-FU, or Carboplatin and Paclitaxel to study whether TAK-676 enhances the localized immune responses compared to both immunotherapy combinations or Carboplatin alone. All investigational drug combinations will be delivered intratumorally in subtherapeutic microdose quantities via the CIVO platform.

The CIVO Microdose Injection Device (MID) penetrates solid tumors and delivers subtherapeutic microdoses of up to eight anti-cancer agents, or combinations of anti-cancer agents, co-injected with CIVO GLO into discrete regions of the tumor. At the time of the planned surgical intervention (4 hours up to four days after the CIVO microdose injection), the injected tumor tissue is then excised and tumor responses are assessed via histological staining of tumor cross-sections sampled perpendicular to each injection column. Co-injection with CIVO GLO enables identification of each injection site during resection as well as in tissues stained for biomarker analysis. Because the platform delivers microdose amounts of each test agent, or combination, directly into the patient's tumor tissue, mechanistic hypotheses can be tested early in the drug development process, consistent with the goals of the 2006 FDA Exploratory Investigational New Drug (IND) Guidance for Industry.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to comply with the study's visit and assessment schedule.
2. Male or female ≥ 18 years of age at Visit 1 (Screening).
3. Pathologic diagnosis of Head and Neck Squamous Cell Carcinoma (HNSCC).
4. Ability and willingness to provide written informed consent. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
5. At least one lesion (primary tumor, recurrent tumor, or effaced metastatic lymph node) ≥ 2 cm in the shortest diameter that is surface accessible for CIVO injection that may be guided by ultrasound if appropriate and for which there is a planned surgical intervention. Treatment plan may include adjuvant radiation or chemotherapy, and patients should have no medical contraindication to surgery.
6. Eastern Cooperative Oncology Group (ECOG) performance score of 0-2.
7. Female patients who:

   * Are postmenopausal for at least one year before the screening visit, OR
   * Are surgically sterile, OR
   * Are of childbearing potential who agree to practice a highly effective method of contraception and one additional effective (barrier) method at the same time (see examples below) from the time of signing the informed consent form (ICF) through four months after the tumor injection procedure OR agree to completely abstain from heterosexual intercourse.

Highly effective methods:

* Intrauterine device (IUD)
* Hormonal (birth control pills/oral contraceptives, injectable contraceptives, contraceptive patches, or contraceptive implants

Other effective methods (barrier methods):

* Latex condom
* Diaphragm with spermicide; Cervical cap; Sponge
* Agree to refrain from donating ova during study participation and up to four months after the tumor injection procedure.

Male patients, even if surgically sterile (i.e., status post-vasectomy), who:

* Agree to practice effective barrier contraception from the time of signing the ICF through four months after the tumor injection procedure OR agree to completely abstain from heterosexual intercourse.
* Agree to refrain from donating sperm during study participation and up to four months after the tumor injection procedure.

Exclusion Criteria:

1. Tumors or effaced nodes that are anticipated by the Investigator to lack a sufficient volume of viable tumor tissue (based on available pre-operative imaging, pre-injection ultrasound imaging, or pathology reports) for CIVO injection due to size, location, necrosis, cysts, excessive stroma, or fibrosis.
2. Patients who have received neoadjuvant therapy associated with the surgical intervention described in Inclusion Criterion #5.
3. Tumors near or involving critical structures for which, in the opinion of the treating clinician, injection would pose undue risk to the patient.
4. Female patients who are:

   * Both lactating and breastfeeding, OR
   * Have a positive β-human chorionic gonadotropin (hCG) pregnancy test at screening verified by the Investigator.
5. Any uncontrolled intercurrent illness, condition, serious medical or psychiatric illness, or circumstance that, in the opinion of the Investigator, could interfere with adherence to the study's procedures or requirements, or otherwise compromise the study's objectives.
6. Patients with a history of concurrent second cancers requiring active, ongoing systemic treatment.
7. Patients with active autoimmune diseases requiring treatment or a known history of uncontrolled autoimmune disorders.
8. Patients with known HIV/AIDS with uncontrolled viral load and cluster of differentiation 4 (CD4) less than 200, a known history of other relevant congenital or acquired immunodeficiencies, or known chronic hepatitis B/C.
9. Patients that have received a live vaccine within 4 weeks of the baseline/screening visit.
10. Use of any of the following ≤ 2 weeks prior to CIVO injection:

    1. Chronic systemic immunosuppressive therapy or corticosteroids. Intranasal, inhaled, topical, or local corticosteroid injections (e.g., intra-articular injection), or steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) are exceptions to this criterion.
    2. Biological response modifiers for treatment of active autoimmune disease.
    3. Hematopoietic growth factors.
11. Patients with prior treatment with other stimulator of interferon genes (STING) agonist/antagonist and toll-like receptor (TLR) agonists, or cell therapies within 2 months of the baseline/screening visit.
12. Patients receiving concurrent systemic therapy (e.g., chemotherapy, targeted agent, or immunotherapy, etc.) or radiation therapy 4 weeks prior to screening through the planned surgical intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Quantification of Cell Death and Immune Cell Biomarkers by immuno-histochemistry (IHC) and In-Situ Hybridization (ISH) | 4 hours - 4 days after microdose injection
  Quantification of biomarker-positive and biomarker-negative cells will be performed within the tumor microenvironment around each of the injection sites in each resected patient sample by IHC and ISH. An aggregate analysis of this quantification may be done across patient samples in each substudy to evaluate trends in tumor response. The biomarkers evaluated may include, but are not limited to, biomarkers for cell death (e.g., cleaved caspase 3), T-cells (e.g., Cluster of Differentiation 3 (CD3), Cluster of Differentiation 8/Granzyme B, Cluster of Differentiation), natural killer (NK)/myeloid cells (e.g., Cluster of Differentiation 56/Granzyme B, Cluster of Differentiation 86, Cluster of Differentiation 68, Cluster of Differentiation 163), and proinflammatory cytokines (e.g., interferon gamma, tumor necrosis factor alpha, interferon gamma-induced protein 10).

SECONDARY OUTCOMES:
Number of Patients with Adverse Events | Up to 28 days after microdose injection
  Relationship of adverse event (AE) to study drug(s) or CIVO device will be determined using an AE Relatedness Grading System

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Jenkins, Study Director — Presage Biosciences Clinical Development
Locations (4):
- United States (4):
  - LSU Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati Health, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gundle KR, Deutsch GB, Goodman HJ, Pollack SM, Thompson MJ, Davis JL, Lee MY, Ramirez DC, Kerwin W, Bertout JA, Grenley MO, Sottero KHW, Beirne E, Frazier J, Dey J, Ellison M, Klinghoffer RA, Maki RG. Multiplexed Evaluation of Microdosed Antineoplastic Agents In Situ in the Tumor Microenvironment of Patients with Soft Tissue Sarcoma. Clin Cancer Res. 2020 Aug 1;26(15):3958-3968. doi: 10.1158/1078-0432.CCR-20-0614. Epub 2020 Apr 16. PMID 32299817
- [Background] Klinghoffer RA, Bahrami SB, Hatton BA, Frazier JP, Moreno-Gonzalez A, Strand AD, Kerwin WS, Casalini JR, Thirstrup DJ, You S, Morris SM, Watts KL, Veiseh M, Grenley MO, Tretyak I, Dey J, Carleton M, Beirne E, Pedro KD, Ditzler SH, Girard EJ, Deckwerth TL, Bertout JA, Meleo KA, Filvaroff EH, Chopra R, Press OW, Olson JM. A technology platform to assess multiple cancer agents simultaneously within a patient's tumor. Sci Transl Med. 2015 Apr 22;7(284):284ra58. doi: 10.1126/scitranslmed.aaa7489. PMID 25904742
- [Background] Frazier JP, Bertout JA, Kerwin WS, Moreno-Gonzalez A, Casalini JR, Grenley MO, Beirne E, Watts KL, Keener A, Thirstrup DJ, Tretyak I, Ditzler SH, Tripp CD, Choy K, Gillings S, Breit MN, Meleo KA, Rizzo V, Herrera CL, Perry JA, Amaravadi RK, Olson JM, Klinghoffer RA. Multidrug Analyses in Patients Distinguish Efficacious Cancer Agents Based on Both Tumor Cell Killing and Immunomodulation. Cancer Res. 2017 Jun 1;77(11):2869-2880. doi: 10.1158/0008-5472.CAN-17-0084. Epub 2017 Mar 31. PMID 28364003
- [Background] Dey J, Kerwin WS, Grenley MO, Casalini JR, Tretyak I, Ditzler SH, Thirstrup DJ, Frazier JP, Pierce DW, Carleton M, Klinghoffer RA. A Platform for Rapid, Quantitative Assessment of Multiple Drug Combinations Simultaneously in Solid Tumors In Vivo. PLoS One. 2016 Jun 30;11(6):e0158617. doi: 10.1371/journal.pone.0158617. eCollection 2016. PMID 27359113
- [Background] Moreno-Gonzalez A, Olson JM, Klinghoffer RA. Predicting responses to chemotherapy in the context that matters - the patient. Mol Cell Oncol. 2015 Jun 10;3(1):e1057315. doi: 10.1080/23723556.2015.1057315. eCollection 2016 Jan. PMID 27308571